CLINICAL TRIAL: NCT04108702
Title: Virtual Reality as a New Therapeutic Tool for Chronic Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of participants
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-01515
Record Dates: First submitted 2019-08-15; First posted 2019-09-30 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VR heart (Experimental)
  Interventions: Device: Virtual reality heart; Other: Standard therapy
- VR control (Sham Comparator)
  Interventions: Device: Virtual reality control; Other: Standard therapy
- Standard control (Active Comparator)
  Interventions: Other: Standard therapy

INTERVENTIONS:
Device: Virtual reality heart — Patients will either sit or stand while wearing a head mounted display (HMD, Oculus Rift). A 360° video, showing a neutral body from the back in a neutral room, will be projected onto the HMD.
  We will record the patients' ECG throughout the entire experiment. Raw data (ECG) are acquired with Arduino and in-house software will detect, in real time, the peak of each R-wave from the recorded ECG data and trigger an additional visual stimulus (e.g. a flashing outline surrounding the virtual body) that flashes on and off SYNCHRONOUSLY with respect to the participant's heartbeat. The silhouette surrounding the virtual body flashes for a duration of 100ms and with a sinusoidal opacity.
  Arms: VR heart
Device: Virtual reality control — Patients will either sit or stand while wearing a head mounted display (HMD, Oculus Rift). A 360° video, showing a neutral body from the back in a neutral room, will be projected onto the HMD.
  We will record the patients' ECG throughout the entire experiment. Raw data (ECG) are acquired with Arduino and in-house software will detect, in real time, the peak of each R-wave from the recorded ECG data and trigger an additional visual stimulus (e.g. a flashing outline surrounding the virtual body) that flashes on and off ASYNCHRONOUSLY with respect to the participant's heartbeat. The silhouette surrounding the virtual body flashes for a duration of 100ms and with a sinusoidal opacity.
  Arms: VR control
Other: Standard therapy — Standard multimodal out-patient therapy program (psychological support, physiotherapy, ergotherapy).

SUMMARY:
Chronic pain is a major health problem and it has been estimate to account for approximately 40% of all medical visits, costing more than $600 billion annually in the United States alone. Given that pharmacological and non-pharmacological treatments for chronic pain are often difficult and may be associated with limiting side effects, technology-based interventions using virtual reality (VR) may be a promising alternative treatment option. Recent findings from cognitive neuroscience show that it is possible to manipulate the body schema and to induce a range of well-controlled illusory bodily experiences by exposing participants to conflicting multisensory bodily inputs using VR, that are associated with changes in pain perception and somatosensory processing in healthy subjects and chronic pain patients. In the current project the investigators plan to follow up on these findings in patients suffering from chronic pain affecting the whole body, e.g. fibromyalgia. The project is planned as a single center clinical study at the Department of Neurology and Psychosomatic Medicine, Inselspital Bern, in cooperation with the Pain Center Inselspital Bern, the Department of Biomedical Engineering; University Bern and the Department of Psychology, University of Bern. The investigators want to explore the analgesic effect of a specific multisensory illusion (e.g. the cardio-visual illusion) in patients suffering from chronic pain as compared to a control condition (single-blinded, randomized clinical trial) using psychometric and algometric methods. Moreover, the investigators would like to assess the physiological changes associated with pain reduction, study the reduction of psychological distress and improved well-being and assess the subjective acceptance of VR as a possible treatment option for patients with chronic pain. Importantly, the investigators plan to develop and test an easy to use, mobile VR setup as a long-term treatment option for patients with chronic pain. Given that chronic pain is a major health problem, the investigators believe that there is a huge market potential for an easy to use, noninvasive and effective treatment option and a possible technology transfer.

ELIGIBILITY:
Inclusion criteria

* A diagnosis of fibromyalgia according to current diagnostic criteria
* Aged > 18 years old
* Capable of judgement
* Willing to participate in the study (by signing the informed consent form)
* Able to follow the study protocol

Exclusion criteria

* Presence of psychosis or major depression with suicidal risk
* History of alcohol or drug abuse
* Inability to follow the procedures of the study, e.g. due to language problems, inability to wear head-mounted display
* Arrythmia, such as atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Pain perception using numeric rating scale VR therapy vs. standard therapy | 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to standard therapy (single-blinded, randomized clinical trial) after 6 weeks using a numeric rating scale (0-10; 0=no pain, 10= max. pain)
Pain perception using patient global impression of change VR therapy vs. standard therapy | 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to standard therapy (single-blinded, randomized clinical trial) after 6 weeks using the Patient global impression of change questionnaire (1-7; 1=very much improved, 7=very much worse).
Pain perception (algometry) VR therapy vs. standard therapy | 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to standard therapy (single-blinded, randomized clinical trial) after 6 weeks using an Algometer:
  The Pain pressure detection threshold to determine hypersensitivity to pain is measured with a standard electronic algometer (Somedic Type II) by bilateral testing on the middle fingers. The electronic algometer is calibrated following the standard protocol as recommended by the manufacturer and set to deliver a steadily increasing pressure (50 kilopascal for 1 s). In this method, the investigators check for the threshold at which non-painful perception of pressure changes to painful perception in response to the gradually increased pressure applied. Low thresholds correspond to high pain sensitivity.
Pain perception (algopeg) VR therapy vs. standard therapy | 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to standard therapy (single-blinded, randomized clinical trial) after 6 weeks using Algopeg:
  The algometric measurement method to detect hyperalgesia will be carried out by means of a pressure pain provocation test. For this type of algometry, we will use a standardized peg with a clamping force of exactly 10 Newton at an extension of 5 mm (Type Algopeg).The pressure is applied on the middle finger and the ear lobes for 10 s each and is invariable. The pegs pressure exerted on an ear lobe is perceived as being consistently and clearly above the pain threshold. The patient indicates the pain intensity on a numerical rating scale (NRS) on which 0 stands for "no pain" and 10 stands for "the most intense pain imaginable". High NRS values correspond with high pain sensitivity/hyperalgesia.

SECONDARY OUTCOMES:
Pain perception (numeric rating scale) VR therapy vs. VR control | 6 weeks and 10 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using Numeric rating scale (0-10; 0=no pain, 10= max. pain).
Pain perception (patient global impression of change) VR therapy vs. VR control | 6 weeks and 10 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using the Patient global impression of change questionnaire (1-7; 1=very much improved, 7=very much worse)
Pain perception (algometric) VR therapy vs. VR control | 6 weeks and 10 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using algometry:
  The Pain pressure detection threshold to determine hypersensitivity to pain is measured with a standard electronic algometer (Somedic Type II) by bilateral testing on the middle fingers. The electronic algometer is calibrated following the standard protocol as recommended by the manufacturer and set to deliver a steadily increasing pressure (50 kilopascal for 1 s). In this method, the investigators check for the threshold at which non-painful perception of pressure changes to painful perception in response to the gradually increased pressure applied. Low thresholds correspond to high pain sensitivity.
Pain perception (algopeg) VR therapy vs. VR control | 6 weeks and 10 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using algopeg:
  The algometric measurement method to detect hyperalgesia will be carried out by means of a pressure pain provocation test. For this type of algometry, we will use a standardized peg with a clamping force of exactly 10 Newton at an extension of 5 mm (Type Algopeg).The pressure is applied on the middle finger and the ear lobes for 10 s each and is invariable. The pegs pressure exerted on an ear lobe is perceived as being consistently and clearly above the pain threshold. The patient indicates the pain intensity on a numerical rating scale (NRS) on which 0 stands for "no pain" and 10 stands for "the most intense pain imaginable". High NRS values correspond with high pain sensitivity/hyperalgesia.
Heart rate variability | During each intervention, up to 6 weeks
  Inter-beat intervals are calculated as the time between two successive R spikes using the ECG signals as acquired during CV stimulation. Raw data are processed in Matlab® (The MathWorks Inc., Natick, USA) with the HRV Analysis Software (HRVAS: HRV Analysis Software). For each subject and each condition, we calculate the square root of the mean squared differences of successive beats intervals (RMSSD), which estimates the short term components of HRV and is commonly used over short recording periods. As HRV pain-related changes occurs mainly in high frequencies (i.e. power spectrum between 0.15 to 0.40 Hz), we then compute frequency-domain HRV analysis and calculated the power spectrum density using Welch's methods for Fast-Fourier Transform.
Hamilton anxiety and and depression scale (HADS) | 6 weeks and 10 weeks
  Study the reduction of psychological distress measured through the Hamilton anxiety and depression scale (Score Anxiety 0-7 normal, 8-10 borderline, 11-21 abnormal; Score depression 0-7 normal, 8-10 borderline, 11-21 abnormal)
Beck depression inventory (BDI II) | 6 weeks and 10 weeks
  Study the reduction of psychological distress measured through the Beck depression inventory. BDI-II contains 21 questions, each answer being scored on a scale value of 0 to 3. Higher total scores indicate more severe depressive symptoms. The standardized cutoffs used are: 0-13: minimal depression; 14-19: mild depression; 20-28: moderate depression; 29-63: severe depression.
WHO 5 Well Being Index | 6 weeks and 10 weeks
  Study well-being through the WHO 5 Well Being Index.
  The WHO-5 consists of five statements, which respondents rate according to the scale below (in relation to the past two weeks).
  All of the time = 5, At no time = 0.
  The total raw score, ranging from 0 to 25, is multiplied by 4 to give the final score, with 0 representing the worst imaginable well-being and 100 representing the best imaginable well-being.
Pain perception (numeric rating scale) | After each intervention, up to 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using the numeric rating scale (0-10; 0=no pain, 10= max. pain).
Pain perception (algometer) | After each intervention, up to 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using algometry:
  The Pain pressure detection threshold to determine hypersensitivity to pain is measured with a standard electronic algometer (Somedic Type II) by bilateral testing on the middle fingers. The electronic algometer is calibrated following the standard protocol as recommended by the manufacturer and set to deliver a steadily increasing pressure (50 kilopascal for 1 s). In this method, the investigators check for the threshold at which non-painful perception of pressure changes to painful perception in response to the gradually increased pressure applied. Low thresholds correspond to high pain sensitivity.
Pain perception (algopeg) | After each intervention, up to 6 weeks
  Explore the analgesic effect of the cardio-visual illusion in patients suffering from chronic pain as compared to a VR control condition using algopeg. The algometric measurement method to detect hyperalgesia will be carried out by means of a pressure pain provocation test. For this type of algometry, we will use a standardized peg with a clamping force of exactly 10 Newton at an extension of 5 mm (Type Algopeg).The pressure is applied on the middle finger and the ear lobes for 10 s each and is invariable. The pegs pressure exerted on an ear lobe is perceived as being consistently and clearly above the pain threshold. The patient indicates the pain intensity on a numerical rating scale (NRS) on which 0 stands for "no pain" and 10 stands for "the most intense pain imaginable". High NRS values correspond with high pain sensitivity/hyperalgesia.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Heydrich, MDPhD, Principal Investigator — Inselspital Bern, University of Bern

IPD SHARING:
Plan to Share IPD: No